CLINICAL TRIAL: NCT05107895
Title: The Effect of Online Coping Skills Training on Stress, Social Problem Solving, and Coping Ways in Youths: A Randomized Controlled Study
Brief Title: The Effect of Online Coping Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esma Ozkan, Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/156
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Coping Skills

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: the researcher who made the initial and final evaluations was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): A 10-week coping skills training was given to the training group from the randomly separated groups. The Coping Skills Training program will take place in a total of 10 online sessions, and the entire program was implemented in 10 weeks. The duration of each session is between 40 and 50 minutes, and it is determined as 5 minutes of introduction to the session, recognizing the general topics, 5 minutes of briefly summarizing the previous session, and the subject of the session for 30-40 minutes. In all sessions, reflections previously prepared with the power point program were used. In the sessions, question-answer method, audio-visual (audio-visual) method, role-playing and performance feedback phases were used when necessary. In addition to knowledge, experiences were also emphasized in education and it was possible to make comparisons with the subject learned in education.
  Interventions: Behavioral: online coping skills training
- Comparator: Control group (Active Comparator): The control group will be informed about their coping skills for a week. Both groups will receive a final evaluation 10 weeks later and a follow-up evaluation 1 month after the last evaluation.
  Interventions: Behavioral: online coping skills training

INTERVENTIONS:
Behavioral: online coping skills training — Young people with high levels of stress were given online coping trainings. The content of this training was primarily aimed at raising awareness about stress by giving information about stress, and then information about coping methods with stress was shared and training on problem solving skills was provided.

SUMMARY:
An announcement will be made on Whatsapp and Instagram social media accounts for the young people who will participate in the research, and preliminary evaluations will be taken from the young people who have stated that they want to participate via e-mail and who meet the working criteria, and randomization will be provided with a computer program. A 10-week coping skills training will be given to the training group from the randomly allocated groups. The control group will be informed about their coping skills for 1 week. Both groups will receive a final evaluation 10 weeks later and a follow-up evaluation 1 month after the last evaluation.

DETAILED DESCRIPTION:
Inclusion criteria

* be over 18 years old
* No barriers to communication
* Not having any health problems
* Getting a score of 11 or higher on the Perceived Stress Scale Exclusion criteria
* Being over 25 years old Being receiving a concurrent psychological treatment/therapy Sample Size 90 participants will be divided into two groups as intervention and control with the online randomization program. It is foreseen that there will be approximately 45 young people in each group.

research design In this study, pretest-posttest and follow-up design including control and training groups will be used.

An announcement will be made on Whatsapp and Instagram social media accounts for the young people who will participate in the research, and preliminary evaluations will be taken from the young people who have stated that they want to participate via e-mail and who meet the working criteria, and randomization will be provided with a computer program. A 10-week coping skills training will be given to the training group from the randomly allocated groups. The control group will be informed about their coping skills for 1 week. Both groups will receive a final evaluation 10 weeks later and a follow-up evaluation 1 month after the last evaluation.

Independent Variables of the Research Coping Skills Training Dependent Variables of the Research Ways of Coping with Stress Scale Perceived Stress Scale (PSS) Social Problem Solving Inventory- Short Form Trait Anxiety Scale Data Collection Tools The data of the research will be obtained with Personal Sociodemographic Information Form, Ways of Coping with Stress Scale, Perceived Stress Scale (PSO) and Social Problem Solving Inventory-Short Form.

Personal Information form: It consists of questions to determine introductory features such as age, gender, marital status, educational status, occupation, health insurance, family structure.

The Ways of Coping Scale, Perceived Stress Scale, Social Problem Solving Inventory-Short Form (SPSI-SF) and Trait Anxiety Scale (STAI-2) will be used in the assessments.

Coping Skills Training

The Coping Skills Training program will take place in a total of 10 sessions, and it is planned to be implemented in a way that the entire program will be completed in 10 weeks. The duration of each session is between 40 and 50 minutes, and it is determined as 5 minutes of introduction to the session, recognizing the general topics, 5 minutes of briefly summarizing the previous session, and the topic of the session for 30-40 minutes. In all sessions, reflections prepared with the power point program will be used. In the sessions, question-answer method, audio-visual (audio-visual) method, role-playing and performance feedback phases will be used when necessary. In addition to knowledge, experiences in education will also be emphasized and it will be possible to make comparisons with the subject learned in education.

SESSION 1: Stress and the concept of stressor SESSION 2: Stress symptoms SESSION 3: Identifying the stressors of the individual, the methods used by the individual, the connection between illness and stress, positive coping methods and recognizing the problem solving steps.

SESSION 4: The effects of stress and stress-related diseases SESSION 5: Asking for help, making a decision SESSION 6: Methods of coping with stress SESSION 7: Problem solving steps SESSION 8: Stress management and therapeutic changes in lifestyle (social support, goal setting) SESSION 9: Examination of breathing techniques SESSION 10: Examining relaxation techniques At the end of the 10th session, the first evaluations will be repeated. Results data will be collected online and automatically entered into a database.

Statistical Method(s) SPSS statistical program will be used in statistical analysis. Frequency and/or mean (X) ± standard deviation (X±SD) values will be given according to the suitability of the socio-demographic characteristics of the individuals with the descriptive data. Values obtained before and after the intervention will be evaluated using the Wilcoxon Paired Test. Statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Young people who scored 11 points or more from the Perceived Stress Scale
* 33 points or more from the State-Trait Anxiety Inventory
* No barriers to communication
* Not having any health problems

Exclusion Criteria:

* older than 25 years of age
* continuing any psychotherapy
* using medication

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | 10 week
  It's developed by Cohen, Kamarck & Mermelste in 1983. In this study, the scale adapted to Turkish was used. A five-point Likert scale (0 not at all, 4 very often) with a score between 11 and 26 indicates a low stress level, between 27 and 41 indicates a medium stress level, and between 42 and 56 indicates a high stress level.

SECONDARY OUTCOMES:
Trait Anxiety Inventory (STAI) | 10 week
  It determines how the individual feels in general, independent of the current situation and conditions. The Trait Anxiety Inventory is a 4-point Likert-type scale: (1) Almost never, (2) Sometimes, (3) Often, and (4) Almost always. The score obtained in the total of the scale takes the values of minimum 20 and maximum 80. A high total score indicates an increase in anxiety, a low score indicates a decrease in anxiety. .
The Scale of Coping Styles with Stress | 10 week
  Developed by Folkman and Lazarus, the scale was shortened by Şahin and Durak (1995). and adapted into Turkish. The evaluation of the items in this scale, which consists of 30 items, is made between 0-3, and the 1st and 9th items are scored by being reversed. There are 5 dimensions in the scale: self-confident approach (7 items), optimistic approach (5 items), helpless approach (8 items), submissive approach (6 items) and seeking social support (4 items). 1995). Minimum score is 0. Maximum score is 90.
Social Problem Solving Inventory-Short Form (SPSI-SF) | 10 week
  consists of two dimensions: "problem orientation" and "problem solving styles". In the problem orientation dimension, there are two subscales: positive problem orientation and negative problem orientation. The problem solving style dimension consists of three subscales: rational problem solving, impulsive/carelessness styles, and avoidance styles. The measurement tool consists of 5 subscales in total. There are 25 items in total in the scale. Items are graded on a five-point scale, from 0 (not at all) to 4 (totally appropriate). inimum score is 0 and maximum score is 100 point.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal information will also be kept confidential by researchers in accordance with the law on the protection of personal information. However, if the journal editor or referees to whom the research is sent want to see the data, it can be shared for information purposes.